CLINICAL TRIAL: NCT01573442
Title: Randomized Double-Blind Placebo Controlled Study of Testosterone in the Adjuvant Treatment of Postmenopausal Women With Aromatase Inhibitor Induced Arthralgias
Brief Title: Testosterone in Treating Postmenopausal Patients With Arthralgia Caused by Adjuvant Aromatase Inhibitor Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A221102; CDR0000730083 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-00719 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA037447 (NIH); UG1CA189823 (NIH)
Record Dates: First submitted 2012-04-06; First posted 2012-04-09 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Arthralgia; Breast Cancer; Hot Flashes; Musculoskeletal Complications; Sexual Dysfunction
Keywords: hot flashes; musculoskeletal complications; sexual dysfunction; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; arthralgia; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Arthralgia; Breast Neoplasms; Hot Flashes; Sexual Dysfunction, Physiological | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive testosterone (0.264mL) topical application daily for six months.
  Interventions: Drug: testosterone
- Arm II (Placebo Comparator): Patients receive placebo (0.264mL) topical application daily for six months.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: testosterone — 10.4 mg
  Arms: Arm I
Other: placebo
  Arms: Arm II

SUMMARY:
This randomized phase III trial studies testosterone to see how well it works compared to placebo in treating postmenopausal patients with arthralgia (joint pain) caused by anastrozole or letrozole. Testosterone may help relieve moderate or severe arthralgia associated with the use of aromatase inhibitors, such as anastrozole or letrozole.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, phase III trial evaluating subcutaneous testosterone for the alleviation of aromatase inhibitor induced arthralgia. A parallel group design will be utilized for this two-arm study: subcutaneous testosterone vs. placebo. Patients are stratified according to baseline pain score (5-6 vs. 7-10) and age (< 50 vs. 50-60 vs. > 60). The primary objective is to determine whether testosterone will reduce AI-induced arthralgia and associated joint symptoms. The secondary objective is to explore whether testosterone will have an acceptable safety and tolerability profile, with particular reference to androgenic adverse events including acne, hirsutism, and alopecia.

Patients are followed up to six months as defined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Receiving anastrozole (1mg) or letrozole (2.5 mg) orally once a day, for ≥ 21 days prior to registration and plan to continue it throughout the duration of study
3. Body Mass Index (BMI) between 18 and 35 kg/m^2
4. Women who have undergone a total mastectomy or breast conserving surgery for primary breast cancer +/-chemo, +/-radiotherapy.
5. Must have BOTH ER and PR receptor-positive tumors and BOTH must be ≥26% positive. Alternatively, if ER and PR are determined by Allred score, the score needs to be 5 or higher
6. Women who are postmenopausal by surgery, radiotherapy or presence of natural amenorrhea ≥ 12 months
7. ≥ 5/10 arthralgia (in hands, wrist, knees, or hips) while being treated with anastrozole or letrozole which is felt by the patient to be caused by their aromatase inhibitor as defined in the protocol. Note: Patients may, or may not, be taking non-opioid analgesics
8. Ability to complete questionnaire(s) by themselves or with assistance
9. ECOG Performance Status (PS) 0, 1 or 2
10. Willing to provide informed written consent
11. Willing to return to an Alliance enrolling institution for follow-up
12. Willing to provide blood samples for correlative research purposes
13. Laboratory values prior to registration as defined in the protocol:

    1. Creatinine ≤1.5 x ULN
    2. Hemoglobin > 11 g/dL
    3. WBC > 3.0
    4. Platelet Count > 100,000
    5. SGOT (AST) ≤ 1.5 x ULN

Exclusion Criteria:

1. Presence of residual or recurrent cancer (locally or metastatic)
2. Diabetes mellitus or glucose intolerance, defined as a fasting glucose >125 mg/dL
3. History of coronary artery disease (angina or myocardial infarction)
4. Patients on hormone replacement therapy (HRT) ≤ 4 weeks prior to registration. This includes the use of vaginal estrogen therapy.
5. Known hypersensitivity to any component of testosterone.
6. Prolonged systemic corticosteroid treatment, except for topical applications (e.g. for rash), inhaled sprays (e.g. for obstructive airway diseases), eye drops or local insertion (e.g. intra-articular). Note: Short duration (< 2 weeks) of systemic corticosteroids is allowed (e.g. for chronic obstructive pulmonary disease) but not within 30 days prior to registration.
7. Receiving any other investigational agent
8. History of a deep venous thrombosis or a thromboembolism
9. Concurrent use of the aromatase inhibitor exemestane, as it is structurally similar to an androgen
10. Concurrent radiation therapy or chemotherapy
11. Current or planned use of cyclosporine, anticoagulants, oxphenbutazone, insulin, oral or injectable vitamin D doses over 4,000IU/day, or tamoxifen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, MD, Study Chair — Mayo Clinic
Locations (529):
- United States (528):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Memorial and Saint Elizabeth's Health Care Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Saint Elizabeth Fort Thomas, Fort Thomas, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Saint Mary's Regional Medical Center, Lewiston, Maine
  - Unspecified Site, Rockville, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Gaston Hematology and Oncology Associates-Belmont, Belmont, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Carolina Surgical Clinic of Charlotte PA, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Gaston Hematology and Oncology Associates, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University Pointe, West Chester, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Kingsport, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Nashville Breast Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - IMG Hematology Oncology 8501, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic Cancer Center - Eau Claire, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Cathcart-Rake E, Novotny P, Leon-Ferre R, Le-Rademacher J, Storrick EM, Adjei AA, Terstriep S, Glaser R, Giuliano A, Mitchell WR, Page S, Austin C, Deming RL, Ferreira MA, Lafky JM, Birrell SN, Loprinzi CL. A randomized, double-blind, placebo-controlled trial of testosterone for treatment of postmenopausal women with aromatase inhibitor-induced arthralgias: Alliance study A221102. Support Care Cancer. 2021 Jan;29(1):387-396. doi: 10.1007/s00520-020-05473-2. Epub 2020 May 6. PMID 32372176
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/about-cancer/treatment/clinical-trials/search/v?id=NCI-2012-00719&q=A221102
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II (Placebo): Patients receive placebo (0.264mL) topical application daily for six months.
- Arm I (Testosterone): Patients receive testosterone (0.264mL) topical application daily for six months.
Period: Overall Study
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Started | 113 | 114
Completed | 104 | 104
Not Completed | 9 | 10
Not completed — Cancels | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm II (Placebo) | Arm I (Testosterone) | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.7) | 59.9 (8.7) | 60.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 104 | 208
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 94 | 100 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 81 | 81 | 162
    1 | 23 | 20 | 43
    2 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Item #3 (Average) of the Brief Pain Inventory (BPI) Average Pain From Baseline to Month 3
Description: The average change in Brief Pain Inventory (BPI) Average Pain scores between baseline and month 3 using Wilcoxon test are reported for each arm below. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: From baseline to 3 months
Population: Patients who completed item #3 (average) of the BPI at baseline and month 3 time points are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 76 | 82
score on a scale | -1.9 (2.5) | -2.0 (2.5)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.4952, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Improvement in BPI Average Pain From Baseline to Month 3
Description: "2. Was there an improvement in BPI Average Pain from baseline to month 3?"
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 104 | 104
Participants
  No | 55 | 45
  Yes | 49 | 59
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.2116, Fisher Exact

3. Primary Outcome: Change in BPI Average Change From Baseline Pain Score to Month Six Average Pain Score
Description: Change in BPI Average Change from Baseline Pain Score to Month Six Average Pain Score. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: Baseline and 6 months
Population: Patients who completed item #3 (average) of the BPI at baseline and month 6 time points are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 68 | 63
score on a scale | -2.2 (2.7) | -1.9 (2.2)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.6760, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in BPI Average Pain From Baseline to Month 1-6
Description: Change in BPI Average Pain from baseline to month 1-6. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: Baseline and months 1-6
Population: Number analyzed below are based on patients who completed the BPI Average Pain item at baseline and specified month.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 104 | 104
score on a scale
  From baseline to month 1: number analyzed (Participants) | 88 | 89
  From baseline to month 1 | -1.2 (2.2) | -1.7 (2.1)
  From baseline to month 2: number analyzed (Participants) | 78 | 77
  From baseline to month 2 | -1.9 (2.3) | -1.9 (2.2)
  From baseline to month 3: number analyzed (Participants) | 76 | 82
  From baseline to month 3 | -1.9 (2.5) | -2.0 (2.5)
  From baseline to month 4: number analyzed (Participants) | 74 | 79
  From baseline to month 4 | -2.1 (2.5) | -2.4 (2.5)
  From baseline to month 5: number analyzed (Participants) | 69 | 73
  From baseline to month 5 | -2.1 (2.7) | -2.0 (2.6)
  From baseline to month 6: number analyzed (Participants) | 66 | 63
  From baseline to month 6 | -2.2 (2.8) | -1.9 (2.2)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); From baseline to month 1; Test type: Superiority; p = 0.029, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm II (Placebo) vs Arm I (Testosterone); From baseline to month 2; Test type: Superiority; p = 0.8214, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm II (Placebo) vs Arm I (Testosterone); From baseline to month 3; Test type: Superiority; p = 0.4952, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Arm II (Placebo) vs Arm I (Testosterone); From baseline to month 4; Test type: Superiority; p = 0.5232, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Arm II (Placebo) vs Arm I (Testosterone); From baseline to month 5; Test type: Superiority; p = 0.5522, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Arm II (Placebo) vs Arm I (Testosterone); From baseline to month 6; Test type: Superiority; p = 0.7005, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With Grade 3 Or Higher Adverse Events Considered At Least Possibly Related to Treatment
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 6 months
Population: Only patients who received at least one cycle of treatment and had adverse events assessed were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 101 | 100
Participants
  grade 3 | 4 | 8
  grade 4 | 1 | 1

6. Secondary Outcome: Number of Patients Who Reported Alopecia Using CTCAE 4.0
Description: The number of patients who reported alopecia using CTCAE 4.0 is reported below for each arm.
Time Frame: Up to 6 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 101 | 100
Participants | 0 | 0

7. Secondary Outcome: Number of Patients Who Reported Acne Using CTCAE 4.0
Description: The number of patients who reported acne using CTCAE 4.0 is reported below for each arm.
Time Frame: Up to 6 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 101 | 100
Participants | 0 | 0

8. Secondary Outcome: Number of Patients Who Reported Hirsutism Using CTCAE 4.0
Description: The number of patients who reported hirsutism using CTCAE 4.0 is reported below for each arm by grade.
Time Frame: Up to 6 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 101 | 100
Participants
  0-None | 94 | 87
  1-Mild | 7 | 10
  2-Moderate | 0 | 3
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.139, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Hot Flash Frequency From Baseline to Week 8
Description: Change in hot flash frequency from baseline to week 8. Hot flash frequency is a count of the number of hot flashes per day and is a number from 0 to infinity. Higher values are worse.
Time Frame: baseline and week 8
Population: Patients who completed the questionnaire at baseline and week 8 are included in this analysis.
Measure: Mean (Standard Deviation); unit: hot flashes/day
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 77 | 72
hot flashes/day | -10.9 (20.6) | -11.4 (19.3)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.8761, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: The Change of Libido From Baseline to Month 3 as Measured by the MENQOL
Description: Change in how bothered are you by decreased sex drive from baseline to month 3. This is assessed using one question off of the MENQOL (Menopause-Specific Quality of Life) questionnaire. The question asks "How bothered are you by a decrease in your sexual drive". This is collected on a scale ranging from 0=Not at all bothered to 6=Extremely bothered, with higher values being worse.
Time Frame: baseline and month 3
Population: Patients who completed MENQOL libido question 'how bothered are you by decreased sex drive' at baseline and month 3 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 104 | 103
score on a scale | -0.5 (2.1) | -1.3 (2.4)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.0176, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: The Change of Menopause Specific Quality of Life From Baseline to Month 3 as Measured by MENQOL "How Bothered Are You by Hot Flashes"
Description: The change of menopause specific quality of life from baseline to month 3 as measured by MENQOL "how bothered are you by Hot Flashes". This is one question from the MENQOL (Menopause-Specific Quality of Life) questionnaire. The question asks "How bothered are you by hot flashes or flushes". This is collected on a scale ranging from 0=Not at all bothered t 6=Extremely bothered, with higher values being worse.
Time Frame: baseline and month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 104 | 104
score on a scale | -1.4 (2.3) | -1.4 (2.4)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.7077, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in BPI Worst Pain From Baseline to Month 3
Description: Change in BPI Worst Pain from baseline to month 3. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: baseline and month 3
Population: Patients who complete the BPI Worst item at baseline and month 3 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 76 | 82
score on a scale | -2.5 (2.7) | -2.4 (2.6)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.8748, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change in BPI Least Pain From Baseline to Month 3
Description: Change in BPI Least Pain from baseline to month 3. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: baseline and month 3
Population: Patients who completed the BPI Least pain item at baseline and month 3 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 76 | 82
score on a scale | -1.0 (2.8) | -1.3 (2.3)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.4335, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change in BPI Pain Right Now From Baseline to Month 3
Description: Change in BPI Pain right now from baseline to month 3. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: baseline and month 3
Population: Patients who completed the BPI pain right now item at baseline and month 3 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 76 | 82
score on a scale | -1.6 (3.0) | -2.1 (2.7)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.286, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change in Average Joint Stiffness From Baseline to Month 3 as Measured by BPI Item #5 (Joint Stiffness)
Description: Change in average joint stiffness from baseline to month 3. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: baseline and month 3
Population: Patients who completed the BPI item #5 on joint stiffness at baseline and month 3 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 76 | 82
score on a scale | -2.0 (2.7) | -2.2 (2.9)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.7694, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: The Intrapatient Change in Activity Level (Interference of Activity) for Each Month From Baseline as Measured by Item#6 (Interference) of the BPI-AIA.
Description: The intrapatient change in activity level (interference of activity) for each month from baseline as measured by item#6 (interference) of the BPI-AIA. Change in general activity from baseline to month 3. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: baseline and month 3
Population: Patients who completed the BPI item #6 at baseline and month 3 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
Number analyzed (Participants) | 78 | 80
score on a scale | -2.1 (3.0) | -2.1 (3.1)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Testosterone); Test type: Superiority; p = 0.9609, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events are assessed ≤ 30 days prior to registration and at the end of Months 3 and 6
Description: Each CTCAE term is a representation of a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who completed at least 1 cycle of tx & AEs were assessed. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Arm II (Placebo) | Arm I (Testosterone)
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/100
Serious Adverse Events (participants affected / at risk) | 1/101 | 5/100
Other Adverse Events (participants affected / at risk) | 23/101 | 25/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm II (Placebo) (N=101) | Arm I (Testosterone) (N=100)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm II (Placebo) (N=101) | Arm I (Testosterone) (N=100)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Hirsutism (Skin and subcutaneous tissue disorders) | 7 (11) | 13 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (12)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT01573442/Prot_SAP_ICF_000.pdf